CLINICAL TRIAL: NCT01140048
Title: An Observational Follow-Up Study of Pediatric Patients Who Participated in a Previous Respiratory Syncytial Virus (RSV)-Induced Bronchiolitis Study of Montelukast
Brief Title: Respiratory Syncytial Virus (RSV) Follow-Up Study (MK-0476-374)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: 0476-374; 2010_026 (Other: Merck Registration ID); MK-0476-374 (Other: Meck Protocol ID)
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Results first posted 2012-10-05 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Respiratory Syncytial Virus Bronchiolitis
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Enrolled Participants: All participants who completed Protocol 272 and were enrolled in Protocol 374

SUMMARY:
This is a prospective, multicenter, observational study in participants who completed the 24-week, placebo-controlled MK-0476 Protocol 272 (NCT00076973) study of montelukast in the treatment of respiratory symptoms subsequent to RSV-induced bronchiolitis. The purpose of this study is to better understand the clinical and demographic correlates of asthma and atopic disorders in children (through the age of 6 years) with a history of severe RSV-induced bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

* successfully completed MK-0476 Protocol 272
* had RSV-induced bronchiolitis at entry into Protocol 272

Exclusion Criteria:

* had developed or had been diagnosed with any illness or congenital disorder that could be immediately life threatening

Ages: 18 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study sample includes participants who completed all visits of Protocol 272 from approximately 38 study sites worldwide. Participants enrolled in Protocol 272 were 3- to 24-month-old children with their first or second episode of "severe" RSV-induced bronchiolitis.
Sampling Method: Non-Probability Sample
Enrollment: 343 (Actual)
Dates: Start 2007-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Lu S, Hartert TV, Everard ML, Giezek H, Nelsen L, Mehta A, Patel H, Knorr B, Reiss TF. Predictors of asthma following severe respiratory syncytial virus (RSV) bronchiolitis in early childhood. Pediatr Pulmonol. 2016 Dec;51(12):1382-1392. doi: 10.1002/ppul.23461. Epub 2016 May 6. PMID 27152482

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Enrolled Participants
Started | 343
Completed | 298
Not Completed | 45
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 13
Not completed — Lost to Follow-up | 31

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 343
Age, Continuous [Mean (Standard Deviation); unit: months] | 45.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143
  Male | 200

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Asthma at 6 Years of Age: Overall and by Prognostic Factor
Description: Asthma was defined as a positive response to the Epidemiology Questionnaire item "Has your child had wheezing or whistling in the chest in the past 6/12 months?" for the period of 12 months prior to age 6 years.
  Prognostic factors for asthma at age 6 years were derived from baseline characteristic, disease characteristic and family history data, and were identified by a forward stepwise regression model.
Time Frame: At 6 years of age
Population: All Enrolled Participants for whom data for the respective Epidemiology Questionnaire item at age 6 years and prognostic factors were available.
Measure: Number; unit: percentage of participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 309
percentage of participants
  With Asthma at Age 6 Years | 6.1
  Relative with Asthma: Yes | 11.2
  Relative with Asthma: No | 3.1
  Gender: Male | 9.6
  Gender: Female | 1.5

2. Secondary Outcome: Percentage of Participants With Atopic Disorders at 6 Years of Age: Overall and by Prognostic Factor
Description: Atopic disorders include allergic rhinitis (AR) and/or atopic dermatitis (AD). Atopic disorders was defined as a positive response to the Epidemiology Questionnaire item "In the past 6/12 months, has your child had a problem with sneezing or runny or blocked nose when he/she did not have a cold or the flu?" for AR and/or a positive response to both of the following items for AD: "Has your child had an itchy rash which was coming and going at any time in the past 6/12 months?" and "Has this itchy rash at any time affected any of the following places: the folds of the elbows, behind the knees, in front of the ankles, under the buttocks, or around the neck, ears, or eyes?" for the period of 12 months prior to age 6 years.
  Prognostic factors for atopic disorders at age 6 years were derived from baseline characteristic, disease characteristic and family history data, and were identified by a forward stepwise regression model.
Time Frame: At 6 years of age
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 309
percentage of participants
  With Atopic Disorders at Age 6 Years | 36.2
  History of AR: Yes | 65.1
  History of AR: No | 25.0
  Relative with Asthma: Yes | 47.4
  Relative with Asthma: No | 29.2

3. Secondary Outcome: Percentage of Participants With Use of Chronic Asthma Therapy at 6 Years of Age: Overall and by Prognostic Factor
Description: Use of Chronic Asthma Therapy for the period of 12 months prior to the age of 6 years was defined by clinical review of reported concomitant medications.
  Prognostic factors for use of chronic asthma therapy at age 6 years were derived from baseline characteristic, disease characteristic and family history data, and were identified by a forward stepwise regression model.
Time Frame: At 6 years of age
Population: All Enrolled Participants for whom data on concomitant asthma therapy at age 6 years and prognostic factors were available.
Measure: Number; unit: percentage of participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 310
percentage of participants
  With Use of Chronic Asthma Therapy at Age 6 Years | 14.5
  History of Asthma: Yes | 32.0
  History of Asthma: No | 6.6
  Region: Africa | 22.5
  Region: Europe | 20.3
  Region: South America | 15.9
  Region: Asia/Pacific | 7.3
  Region: North & Central America | 5.7

ADVERSE EVENTS:
Time Frame: Serious adverse events that occurred within 24 hours following a study procedure
Description: Only serious adverse events related to study-defined procedures that occurred within 24 hours following the procedure were to be reported. Information on non-serious adverse events was not to be collected.
Arm/Group | All Enrolled Participants
Serious Adverse Events (participants affected / at risk) | 0/343
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.